CLINICAL TRIAL: NCT05232097
Title: Behavioral Therapy in Patients With Rumination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jari Punkkinen, Chief, Division of Gastroenterology, Hyvinkää Hospital, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS/23/2022; HUS/2118/2021 (Other: HUCS Ethics Committee)
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Behavior Therapy; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral therapy (Experimental): Behavioral therapy consisting of diaphragmatic breathing exercises and physiotherapy to relax tensed abdominal and thoracic muscles
  Interventions: Behavioral: Behavioral therapy; Behavioral: Physiotherapy

INTERVENTIONS:
Behavioral: Behavioral therapy — Diaphragmatic breathing exercises
Behavioral: Physiotherapy — Body awareness aiming at the patient becoming aware of the tensed thoracic and abdominal muscles and to reduce the tension by relaxation exercises taught by the psychophysical physiotherapist

SUMMARY:
The study aim is to diagnose patients with the rumination syndrome defined by the Rome IV criteria and to treat them with behavioral therapy consisting of diaphragmatic breathing exercises and physiotherapy to relax tensed abdominal and thoracic muscles.

Before referral to the study, gastroscopy, esophageal hgh-resolution manometry and 24-hour esophageal pH and impedance monitoring are required to rule out other esophageal conditions.

Twenty Finnish speaking, 15-70 years old patients will be enrolled in this open study. All patients will visit the gastroenterologist at onset of the study and at 6 months. All patients will be referred to the speech therapist for five one-hour sessions consisting of diaphragmatic belching exercises and to the physiotherapist for two one-hour sessions consisting of exercises to relax tensed thoracic and abdominal muscles. All patients will also visit once the psychologist and dietician.

Symptoms will be evaluated by the Rome IV questionnaire for adult functional gastrointestinal diseases at onset and at the 6-month control. Health-related quality of life, depression, anxiety, functional capacity will be evaluated by specific questionnaires at onset of the study and at the 6-month control. Esophageal high-resolution manometry will be performed at the 6-month control.

DETAILED DESCRIPTION:
Background: Rumination is a subconscious but a volitional, behavioral disorder. Contraction of the abdominal muscles results in an increase of abdominal pressure and a subsequent regurgitation of recently ingested food, followed by rechewing, reswallowing or spitting (1). The diagnosis is based on the Rome IV criteria for functional gastrointestinal disorders and esophageal high-resolution manometry (1, 2). Behavioral therapy consisting of diaphragmatic breathing exercises has proven efficient in these patients (3, 4). Psychophysical physiotherapy was effective in a published patient case (5).

Aim: The study aim is to diagnose patients with rumination syndrome defined by the Rome IV criteria and to treat them with behavioral therapy. The primary aim is a reduction of two points ore more in the rumination frequency measured by the Rome IV questionnaire for adult functional gastrointestinal diseases (6). Secondary aims are improved esophageal high-resolution manometry, health-related quality of life, and functional capacity and reduced anxiety and depression scores.

Patients: 20 Finnish speaking, 15-70 years old patients with rumination symptoms fulfilling the Rome IV criteria will be enrolled in this open study. Before referral to Helsinki University Central Hospital, gastroscopy, esophageal high-resolution manometry and esophageal 24-hour pH and impedance monitoring are required. Adolescents of 15 to 17 years old are referred to the childrens' gastroenterologist and adults 18 years or older are referred to the gastroenterologist. The inclusion criteria consist of rumination symtoms fulfilling the Rome IV criteria but esophageal high-resolution manometry may be negative because rumination cannot be always provoked during the study.The exclusion criteria comprise eating disorder, BMI <14, pregnancy, cognitive or other disorder that disallows behavioral therapy

Methods: Symptoms will be evaluated by the Rome IV questionnaire for adult functional gastrointestinal diseases in all patients. Health-related quality of life will be evaluated by 15D, a 15-dimensional measure of health-related quality of life, depression by Beck Depression Inventory (BDI), anxiety by the Beck Anxiety Inventory (BAI), and functional capacity by WHODAS 2.0, World Health Organization disability assesment schedule 2.0 in the patients 18 years or older (7-10). In the patients 15-17 years old, health-related qualiy of life will be evaluated by 16D, a sixteen-dimensional health-related measure for adolescents (11). All questionnaires will be carried out at the onset of the study and at the 6-month control. Esophageal high-resolution manometry will be performed at the 6-month control.

After the baseline visit to the gastroenterologist, patients will be sent to the speech therapist for five, one-hour sessions consisting of diaphragmatic breathing exercises and to a psychophysical physiotherapist for two one-hours sessions aiming at body-awareness to sense tensed thoracic and abdominal muscles and to relax them through guided exercises. Patients will continue these exercises at home during meals. All patient l visit the psychologist and dietician once to rule out eating disorders and other psychopathological conditions and will be referred to the psychiatrist when necessary. Esophageal high-resolution manometry will be performed at the 6-month control.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV criteria for rumination syndrome fulfilled
* gastroscopy, esophageal HR-manometry and 24-hour pH-impedance monitoring performed before referral to study

Exclusion Criteria:

* eating disorder, BMI <14, pregnancy, cognitive or other disorder that disallows behavioral therapy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jari Punkkinen, Dr, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Helsinki University Hospital, Childrens' Hospital, Helsinki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halland M, Pandolfino J, Barba E. Diagnosis and Treatment of Rumination Syndrome. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1549-1555. doi: 10.1016/j.cgh.2018.05.049. Epub 2018 Jun 12. PMID 29902642
- [Background] Kessing BF, Bredenoord AJ, Smout AJ. Objective manometric criteria for the rumination syndrome. Am J Gastroenterol. 2014 Jan;109(1):52-9. doi: 10.1038/ajg.2013.428. Epub 2013 Dec 24. PMID 24366235
- [Background] Barba E, Accarino A, Soldevilla A, Malagelada JR, Azpiroz F. Randomized, Placebo-Controlled Trial of Biofeedback for the Treatment of Rumination. Am J Gastroenterol. 2016 Jul;111(7):1007-13. doi: 10.1038/ajg.2016.197. Epub 2016 May 17. PMID 27185077
- [Background] Halland M, Parthasarathy G, Bharucha AE, Katzka DA. Diaphragmatic breathing for rumination syndrome: efficacy and mechanisms of action. Neurogastroenterol Motil. 2016 Mar;28(3):384-91. doi: 10.1111/nmo.12737. Epub 2015 Dec 10. PMID 26661735
- [Background] Muurinen T, Walamies M. [Rumination in a young woman]. Duodecim. 2015;131(1):76-9. Finnish. PMID 26245059
- [Background] Palsson OS, Whitehead WE, van Tilburg MA, Chang L, Chey W, Crowell MD, Keefer L, Lembo AJ, Parkman HP, Rao SS, Sperber A, Spiegel B, Tack J, Vanner S, Walker LS, Whorwell P, Yang Y. Rome IV Diagnostic Questionnaires and Tables for Investigators and Clinicians. Gastroenterology. 2016 Feb 13:S0016-5085(16)00180-3. doi: 10.1053/j.gastro.2016.02.014. Online ahead of print. PMID 27144634
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Leyfer OT, Ruberg JL, Woodruff-Borden J. Examination of the utility of the Beck Anxiety Inventory and its factors as a screener for anxiety disorders. J Anxiety Disord. 2006;20(4):444-58. doi: 10.1016/j.janxdis.2005.05.004. Epub 2005 Jul 6. PMID 16005177
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Federici S, Bracalenti M, Meloni F, Luciano JV. World Health Organization disability assessment schedule 2.0: An international systematic review. Disabil Rehabil. 2017 Nov;39(23):2347-2380. doi: 10.1080/09638288.2016.1223177. Epub 2016 Nov 7. PMID 27820966
- [Background] Apajasalo M, Sintonen H, Holmberg C, Sinkkonen J, Aalberg V, Pihko H, Siimes MA, Kaitila I, Makela A, Rantakari K, Anttila R, Rautonen J. Quality of life in early adolescence: a sixteen-dimensional health-related measure (16D). Qual Life Res. 1996 Apr;5(2):205-11. doi: 10.1007/BF00434742. PMID 8998489

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Therapy: Behavioral therapy consisting of diaphragmatic breathing exercises and physiotherapy to relax tensed abdominal and thoracic muscles
  Behavioral therapy: Diaphragmatic breathing exercises
  Physiotherapy: Body awareness aiming at the patient becoming aware of the tensed thoracic and abdominal muscles and to reduce the tension by relaxation exercises taught by the body-mind orientated physiotherapist
Period: Overall Study
Arm/Group | Behavioral Therapy
Started | 11
Completed | 10
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 38 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Finland | 11
Rumination score (self-perceived rumination frequency) [Median (Inter-Quartile Range); unit: units on a scale] — Rumination score measured by question 32 of the Rome 4 diagnostic questionnaire for adult functional gastrointestinal disorders. The question scores the rumination frequency as follows: "In the last 3 months, how often did food come back up into your mouth after you swallowed it ?, 0 = never, 1= fewer than 1 day a month, 2 = 1 day a month, 3 = 2-3 days a month, 4 = 1 day a week, 5 = 2-3 days a week, 6 = most days, 7 = every day, 8 = multiple times per day or all the time".
  units on a scale | 6.5 [5 to 8]
Anxiety score (BAI) [Median (Inter-Quartile Range); unit: Units on a score] — Beck Anxiety Inventory (BAI) Score. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
  Units on a score | 18 [5 to 29]
Depression score (BDI) [Median (Inter-Quartile Range); unit: Score on scale] — Beck Depression Inventory (BDI) Score, scale 0-63. Total score of 0-13 is considered minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
  Score on scale | 12 [6 to 13]
Healt-related quality of life (15D) [Mean (Standard Deviation); unit: units on a scale] — The 15-dimensional measure of health-related quality of life (15D) includes 15 dimensions: breathing, mental function, speech, vision, mobility, usual activities, vitality, hearing, eating, elimination, sleeping, distress, discomfort and symptoms, sexual activity, and depression, each scored from 1 (best possible) to 0 (worst possible). The 15D score, a single index number over all the dimensions, is calculated with the maximum score 1 (no problems on any dimension) and the minimum score 0 (being dead).
  units on a scale | 0.793 (0.171)
Functional capacity (WHODAS 2.0) [Median (Inter-Quartile Range); unit: units on a scale] — The World Health Organization disability assessment schedule 2.0 (WHODAS 2.0) produces domain-specific scores for six different functioning domains -cognition, mobility, self-care, getting along, life activities (household and work) and participation. Each domain is scored from 0 (no disability) to 100 (full disability). The summary score is converted into a metric ranging from 0 to 100, where 0 = no disability and 100 = full disability.
  units on a scale | 26 [7 to 47]
Weight [Median (Inter-Quartile Range); unit: kilograms] — Weigth in kilograms
  kilograms | 71 [51 to 92]

OUTCOME MEASURES:

1. Primary Outcome: Rumination Score (Self-perceived Rumination Frequency)
Description: Rumination score measured by question 32 of the Rome 4 diagnostic questionnaire for adult functional gastrointestinal disorders. The question scores the rumination frequency as follows: "In the last 3 months, how often did food come back up into your mouth after you swallowed it ?, 0 = never, 1= fewer than 1 day a month, 2 = 1 day a month, 3 = 2-3 days a month, 4 = 1 day a week, 5 = 2-3 days a week, 6 = most days, 7 = every day, 8 = multiple times per day or all the time". Scale 0-8, the highest score indicating highest frequency of rumination.
Time Frame: 6-month control
Population: The 10 patients who finished the study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 10
score on a scale | 4 [3 to 5]
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis: the median of differences of the rumination score before and after therapy equals 0; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Patients With Abdominal Pressure Peaks of an Amplitude of 30 mmHg or Higher
Description: Number of patients with abdominal pressure peaks of an amplitude of 30 mm Hg or higher measured by means of esophageal high-reselution manometry indicating rumination.
Time Frame: 6-month control
Population: The 9 patients who were performed manometry at the 6-month control. Out of the 10 patients who finished the study, one refused.
Measure: Count of Participants; unit: Participants
Groups:
- Behavioral Therapy: Behavioral therapy consisting of diaphragmatic breathing exercises and physiotherapy to relax tensed abdominal and thoracic muscles
  Behavioral therapy: Diaphragmatic breathing exercises
  Physiotherapy: Body awareness aiming at the patient becoming aware of the tensed thoracic and abdominal muscles and to reduce the tension by relaxation exercises taught by the body-mind orientated physiotherapist
  Eleven (11) patients participated in the study. One patient was withdrawn from the study because of severe anxiety by doctor´s decision.
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 9
Participants | 6
Statistical Analysis 1: Comparison: Behavioral Therapy; The null hypothesis is that the same number of patients has intragastric pressure peaks indicating rumination before and after therapy; Test type: Other; p = 0.11, Chi-squared

3. Secondary Outcome: Health-related Quality of Life (15D)
Description: The 15D, a 15-dimensional measure of health-related quality of life includes 15 dimensions: breathing, mental function, speech, vision, mobility, usual activities, vitality, hearing, eating, elimination, sleeping, distress, discomfort and symptoms, sexual activity, and depression, each scored from 1 (best possible) to 0 (worst possible). The 15D score, a single index number calculated over all the dimensions, is ranged from the maximum score 1 (no problems on any dimension) to the minimum score 0 (being dead).
Time Frame: 6-month control
Population: The 8 patients who returned the 15D-questionnaire both at baseline and at the 6-month control. Out of the 10 patients who finished the study, 2 did not return the questionnaire at the 6-month control.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 8
units on a scale | 0.845 (0.141)
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis: The differences of means of 15D before and after therapy equals 0; Test type: Other; p = 0.060, t-test, 2 sided

4. Secondary Outcome: Functional Capacity (WHODAS 2.)
Description: WHODAS 2.0, the WHO Disability Assessment Schedule 2.0 questionnaire, covers six domains of functioning, including: Cognition - understanding & communicating, Mobility- moving & getting around, Self-care- hygiene, dressing, eating & staying alone, Getting along- interacting with other people, Life activities- domestic responsibilities, leisure, work & school, and Participation- joining in community activities. Each domain is ranged from 0 (no disability) to 100 (full disability).
  The WHODAS 2.0 summary score consisting of all six domains is converted to metric ranging from 0 to 100, with 0 indicating no disability and 100 full disability.
Time Frame: 6-month control
Population: The 8 patients who returned the WHODAS 2.0 questionnaire both at baseline and at the 6-month control. Out of the 10 patients who finished the study, 2 patients did not return the questionnaire at the 6-month control.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 8
units on a scale | 11 [7 to 26]
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis: The median of differences of WHODAS 2.0 before and after therapy equals 0; Test type: Other; p = 0.865, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Depression Score (BDI)
Description: Beck Depression Inventory (BDI) Score, scale 0-63. Total score of 0-13 is considered minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Time Frame: 6-month control
Population: The 8 patients who returned the BDI-questionnaire both at baseline and at the 6-month control. Out of the 10 patients who finished the study, 2 did not return the questionnaire at the 6-month control.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 8
score on a scale | 7 [4 to 8]
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis : the differences of median BDI before and after behavioral therapy equals 0; Test type: Other; p = 0.149, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Anxiety Score (BAI)
Description: Beck Anxiety Inventory (BAI) Score, scale 0-63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Time Frame: 6-month control
Population: The 8 patients who returned the BAI questionnaire both at baseline and at the 6-month control. Out of the 10 patients who finished the study, 2 did not return the questionnaire at the 6-month control.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 8
score on a scale | 15 [7 to 27]
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis: The differences of median of BAI before and after behavioral therapy equals 0; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Weight
Description: Weight in kilograms
Time Frame: 6-month control
Population: All 10 patients who finished the study.
Measure: Median (Inter-Quartile Range); unit: kilogram
Arm/Group | Behavioral Therapy
Number analyzed (Participants) | 10
kilogram | 71 [56 to 93]
Statistical Analysis 1: Comparison: Behavioral Therapy; Null hypothesis: The differences of median weight before and after therapy equals 0; Test type: Other; p = 0.102, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not assessed systematically but possible arverse effects were registered at the 6-month control.
Groups:
- Behavioral Therapy: Behavioral therapy consisting of diaphragmatic breathing exercises and physiotherapy to relax tensed abdominal and thoracic muscles
  Behavioral therapy: Diaphragmatic breathing exercises
  Physiotherapy: Body awareness aiming at the patient becoming aware of the tensed thoracic and abdominal muscles and to reduce the tension by relaxation exercises taught by the psychophysical physiotherapist
  Eleven (11) patients participated in the study. One patient was withdrawn from the study because of severe anxiety by doctor´s decision.
Arm/Group | Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The patient sample is very small, although we actively recruited patients for two years from the Helsinki University Central Hospital area covering 1.7 million people. This was an open study without any control group, but it would have been both difficult to create an alternative therapy for randomization and unethical given that the patients had difficult rumination occurring most days of the week.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05232097/Prot_SAP_000.pdf